CLINICAL TRIAL: NCT03311945
Title: Phase 3b, Single Arm, Single Site Simplification Study of HIV-1 Infected Patients With Virological Suppression Under the Combination of Lamivudine (150 mg BID) Plus Raltegravir (400 mg BID) Switching to Lamivudine (300 mg QD) Plus Raltegravir (1200 mg QD) : Roll-over Study of the RALAM Clinical Trial (NCT02284035)
Brief Title: Simplification Study of HIV-1 Infected Patients With Virological Suppression Under the Combination of Lamivudine (150 mg BID) Plus Raltegravir (400 mg BID) Switching to Lamivudine (300 mg QD) Plus Raltegravir (1200 mg QD) : Roll-over Study of the RALAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Judit Pich (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor-Investigator, Judit Pich, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RALAM-Roll Over; 2017-000986-60 (EudraCT Number)
Record Dates: First submitted 2017-09-29; First posted 2017-10-17 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections; HIV-1-infection; HIV Seropositivity
Keywords: Raltegravir; Lamivudine
MeSH Terms: conditions — HIV Infections; HIV Seropositivity | interventions — Raltegravir Potassium; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raltegravir + Lamivudine (Experimental): Lamivudine (300 mg QD) plusRaltegravir (1200 mg QD)
  Interventions: Drug: Raltegravir; Drug: Lamivudine

INTERVENTIONS:
Drug: Raltegravir — Raltegravir (1200 mg QD)
Drug: Lamivudine — Lamivudine (300 mg QD)

SUMMARY:
Phase 3b, single arm, single site simplification study of HIV-1 infected patients with virological suppression under the combination of Lamivudine (150 mg BID) plus Raltegravir (400 mg BID) switching to Lamivudine (300 mg QD) plus Raltegravir (1200 mg QD): Roll-over study of the RALAM clinical trial (NCT02284035)

ELIGIBILITY:
Inclusion Criteria:

* Patients in the switch arm who have completed the 24-week follow-up of RALAM (NCT02284035) study and remain virologically suppressed (viral load <50 copies/mL) on dual therapy with lamivudine plus Raltegravir
* Patients who have signed informed consent to participate in the study.

Exclusion Criteria:

* Pregnancy, lactation, or planned pregnancy during the study period
* Any disease or history of disease which, in opinion of the investigator, might confound the results of the study or pose additional risk to patient treatment
* Hepatitis B co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic i Provincial de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All trial subjects were recruited at a single site in Spain: Hospital Clínic de Barcelona. The subjects were patients in the switch arm who completed the 24-week follow-up of RALAM (NCT02284035) study and remained virologically suppressed (viral load <50 copies/mL) on dual therapy with 3TC plus Raltegravir.
  Recruitment start period: 02-May-2018.
Pre-assignment Details: Selection and baseline will be done in the same visit. Performed at Week 0. During this visit, written informed consent was obtained from each patient, and demographic data, medical history, complete physical examination, and laboratory tests (including hematology, biochemistry, and plasma viral load) were performed to confirm eligibility.
Groups:
- RAL+3TC: Lamivudine (300 mg QD) plus Raltegravir (1200 mg QD)
Period: Overall Study
Arm/Group | RAL+3TC
Started | 33
Completed | 30
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir + Lamivudine
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Therapeutic Failure
Description: Proportion of patients that at least present one of the following events: virological failure, change in antirretroviral treatment for any reason, consent withdrawal, loss to follow-up or death.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Raltegravir + Lamivudine: Lamivudine (300 mg QD) plus Raltegravir (1200 mg QD)
Arm/Group | Raltegravir + Lamivudine
Number analyzed (Participants) | 33
Participants
  Patients with therapeutic failure | 3
  Patients without therapeutic failure | 30
Statistical Analysis 1: Comparison: Raltegravir + Lamivudine; Test type: Other; This was a single-arm study without a comparator group; therefore, no formal hypothesis testing was conducted. The primary endpoint-therapeutic failure at 48 weeks-was analyzed descriptively. The proportion of participants experiencing therapeutic failure was calculated for both the intention-to-treat (ITT) and on-treatment (OT) populations. Exact binomial (Clopper-Pearson) 95% confidence intervals were used to estimate the failure rates

2. Secondary Outcome: Change From Baseline in Peripheral Mononuclear Blood Cells HIV-1 Reservoir
Time Frame: 48 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Changes From Baseline in Cholesterol Total
Time Frame: 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Changes From Baseline in Cholesterol LDL
Time Frame: 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Changes From Baseline in Cholesterol HDL
Time Frame: 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Changes From Baseline in Triglycerides
Time Frame: 24 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Changes From Baseline in Insulin Resistance (HOMA-IR)
Time Frame: 24 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in Lumbar and Femoral Bone Mineral Density
Time Frame: 48 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in Plasma 25-OH Vitamin D Levels
Time Frame: 48 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in Urine Beta-2-microglobulin
Time Frame: 48 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (Chronic Kidney Disease Epidemiology CollaborationI)
Time Frame: 48 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Change From Baseline in Urine Protein/Creatinine Ratio
Time Frame: 48 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Changes From Baseline in Biomarkers of Inflammation IL-6
Time Frame: 48 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Changes From Baseline in Biomarker of Mononuclear Activation SD-163
Time Frame: 48 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Changes From Baseline in Biomarker of Mononuclear Activation SD-14
Time Frame: 48 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Changes From Baseline in Biomarker of Inflammation High Sensitivity C-reactive Protein
Time Frame: 48 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Changes From Baseline in Sleep Quality (Pittsburgh Sleep Quality Index) at
Time Frame: 48 weeks
Reporting Status: Not Posted

18. Secondary Outcome: Change From Baseline in EQ-5D-5L
Time Frame: 48 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Incidence of Adverse Events
Time Frame: 48 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Viral Load
Description: Proportion of patients with viral load below ultrasensitive HIV-1 RNA detection limit (limit of detection 1 copy/mL) at 48 weeks
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: Adverse events were assessed systematically at each study visit through clinical evaluation, laboratory testing, and patient self-reporting. Investigators used open-ended questioning, physical examination, and review of laboratory results to detect AEs. Severity was graded using the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. All AEs were recorded in the case report form, including onset, duration, severity, causality, and outcome.
Arm/Group | Raltegravir + Lamivudine
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 16/33
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir + Lamivudine (N=33)
Gastrointestinal (Gastrointestinal disorders) | 9 (9)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dermatological (Skin and subcutaneous tissue disorders) | 2 (2)
Genitourinary (Renal and urinary disorders) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Endocrine (Endocrine disorders) | 1 (1)
Infections (Immune system disorders) | 1 (1)
Systemic (General disorders) | 8 (8) — Affecting more than ne organ or system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT03311945/Prot_SAP_000.pdf